CLINICAL TRIAL: NCT03828916
Title: Single Arm Clinical Evaluation of the Safety and Efficacy of the NuShield® Allograft for Peroneal Tendon Repair
Brief Title: NuShield in Surgical Peroneal Tendon Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NuTech Medical, Inc (Industry)
Collaborators: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2018-01-01
Record Dates: First submitted 2018-07-20; First posted 2019-02-04 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Tendon Injuries; Tendinopathy
Keywords: Tendon Surgery; NuShield
MeSH Terms: conditions — Tendon Injuries; Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NuShield (Other)
  Interventions: Other: NuShield

INTERVENTIONS:
Other: NuShield — SOC surgery with the addition of NuShield

SUMMARY:
The purpose of this study is to evaluate the use of NuShield in subjects requiring surgical tendon repair.

DETAILED DESCRIPTION:
The objective of this clinical trial is to evaluate both the safety and efficacy of using the NuShield® allograft in addition to standard of care surgical procedures in subjects requiring surgical repair of the peroneal tendon. The effects of this treatment will be assessed using:

* Questionnaires

  * Visual Analog Scale Foot and Ankle (VAS FA)
  * FAAM Sport
  * PROMIS Global Health SF
  * Tegner Activity Scale
  * Foot and Ankle Outcomes Instrument (Q1, Q2)
* Swelling assessments
* Ultrasound imaging for tendon thickness, gliding and adhesion formation

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 60 inclusive
* If female, actively practicing a medically relevant method of contraception, abstinent, surgically sterile, or post-menopausal (defined as no menses for at least 12 months)
* Have a diagnosis of one of the following in relation to the peroneal tendon:

  * Tendonitis with MRI confirmation
  * Synovial inflammation
  * Tear
* Diagnosis resulting from acute injury to the tendon

Exclusion Criteria:

* BMI equal to or greater than 35
* Prior injury to the peroneal tendon
* Collagen disorders
* Inflammatory arteriopathies
* Immune compromised
* Diabetic
* Less than 6 months between injury and proposed surgery date
* Steroid injection within the past 6 weeks localized to the treatment area
* Pregnant within the past six (6) months, breast feeding and/or desire to become pregnant during the course of the study, as verified by urine pregnancy test within one week prior to treatment
* History of more than two (2) weeks treatment with immuno-suppressants, including systemic corticosteroids or cytotoxic chemotherapy within one month prior to initial screening, or have received such medications during the screening period, or are anticipated to require such medications during the course of the study
* Taking any investigational drug(s) or therapeutic device(s) within 30 days preceding screening
* History of radiation therapy of the affected foot
* Known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV
* Currently involved in medical litigation, including Worker's Compensation claims of any type
* Unable to understand the objectives of the trial
* Presence of any condition(s) which, in the opinion of the investigator, would compromise the subject's ability to complete this study
* Having a known history of poor adherence with medical treatment
* Express an unwillingness to receive human allograft tissue

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
VAS Foot and Ankle Pain | 6 Months
  Visual Analogue Scale (VAS) foot and ankle pain. Change in pain intensity scores from baseline. VAS is measured in mm (scale 0-100); with 0 indicating worse outcomes and 100 indicating better outcome
FAAM Sports Subscale | 6 Months
  Foot and Ankle Ability Measure (FAAM) Sports Subscale. Changes in FAAM Sport scores from baseline (scale 0-4); with 0 indicating better outcomes and 4 indicating worse outcomes

SECONDARY OUTCOMES:
Adverse Events | up to 1 year
  Evaluations of safety will include serious adverse events or observed and/or volunteered adverse events.
Swelling assessment by investigator | 6 and 12 months
  Circumferential measurement of the limbs. Change in swelling measured in cm
PROMIS Global Health Subscale | 6 and 12 months
  PROMIS® (Patient-Reported Outcomes Measurement Information System) Global Health Subscale. Changes from baseline (scale 1-5); with 5 indicating better outcomes and 1 indicating worse outcomes
Tegner Activity Scale | 6 and 12 months
  Tegner Activity Scale (scale 0-10). Changes from baseline; with 0 indicating worse outcomes and 10 indicating better outcomes
Foot and Ankle Outcome Instrument, Questions 1 and 2 (subscale) | 6 and 12 months
  Patient reported outcome (PRO) measurement of stiffness and swelling (1-5); with 1 indicating better outcomes and 5 indicating worse outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Central Research Associates, Inc., Birmingham, Alabama
  - University of Colorado Health Orthopedics Clinic - Anschutz Medical Campus, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No